CLINICAL TRIAL: NCT04432025
Title: Medication Following Bariatric Surgery for Type 2 Diabetes Mellitus
Acronym: BY-PLUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20HH5928
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: obesity; type 2 diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to the control arm (bariatric surgery- either RYGB or SG) or intervention (bariatric surgery- either RYGB or SG + goal directed medical therapy for t2DM)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients will undergo bariatric surgery- either roux en y gastric bypass or sleeve gastrectomy. Long term diabetes care will be under the supervision of their primary care provider/general practitioner
  Interventions: Procedure: Bariatric surgery
- Intervention (Experimental): Patients will undergo bariatric surgery- either roux en y gastric bypass or sleeve gastrectomy and will have ongoing goal directed medical treatment for their T2DM, titrated to specific end points for BP, HbA1c and lipids.
  Interventions: Procedure: Bariatric surgery + goal directed medical therapy

INTERVENTIONS:
Procedure: Bariatric surgery + goal directed medical therapy — Patients will undergo bariatric surgery (RYGB or SG) with goal directed medical therapy titrated to specific end points for BP, HbA1c and lipids
  Arms: Intervention
Procedure: Bariatric surgery — Patients will undergo bariatric surgery (RYGB or SG) with usual care for diabetes mellitus undertaken by their primary care provider/general practitioner
  Arms: Control

SUMMARY:
The aim of this study is to investigate the continued usage of standard diabetes medications in the post operative period following bariatric surgery to determine whether this approach may improve long term diabetes control. At present, the standard of treatment in patients with type 2 diabetes is that all medication is stopped in the immediate postoperative period and only re-started if symptoms of diabetes re-emerge. Although a large proportion of patients with diabetes will initially go in to remission, 80% experience relapse within five years. This study is needed to determine whether continuing medications is not only safe but will improve long term outcomes for patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* eligible for bariatric surgery according to NICE guidelines (GC 189)
* Type 2 diabetes mellitus
* BMI >30kg/m2

Exclusion Criteria:

* Recent hospitalisation in the past 30 days
* Recurrent hypoglycaemic episodes
* Recurrent hypotensive episodes
* Contraindications to bariatric surgery
* Previous bariatric surgery
* Current pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in each group reaching the composite end point | 5 years
  BP<130/80, HbA1c<6.5%, LDL<2.6mmol/L
Proportion of patients reaching end point for glycemic control | 1 year
  HbA1c<6.5%

SECONDARY OUTCOMES:
Change in body weight | 5 years
  Change in body weight from baseline (kg)
Change in BMI | 5 years
  Change in BMI from baseline (kg/m2)
Change in waist circumference | 5 years
  Change in waist circumference (cm)
Change in lipid control | 5 years
  Proportion of patients achieving good lipid control (LDL<2.6mmol/L)
Change in glycaemic control | 5 years
  Change in long term glycaemic control(HbA1c)
Change in blood pressure | 5 years
  Proportion of patients achieving BP<130/80mmHg
Change in liver function | 5 years
  Proportion of patients achieving normal liver function tests (ALT, GGT, ALP, AST)
Change in renal function | 5 years
  Proportion of patients with normal renal function (plasma Cr, eGFR)
Change in inflammatory markers | 5 years
  Reduction in CRP
Change in urine albumin: creatinine ratio | 5 years
  Proportion of patients in each group with a uACR<30
Change in quality of life | 5 years
  Quality of life change as determined by SF-36 and MPH-H

CONTACTS AND LOCATIONS:
Locations (1):
- University College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
The authors shall make data available to the scientific community with as few restrictions as feasible, ensuring anonymisation, while retaining exclusive use until the publication of major outputs.
Supporting Information: Study Protocol
Time Frame: 6 months
Access Criteria: Free access

REFERENCES:
- [Derived] Sudlow A, Miras AD, Cohen RV, Kahal H, Townley J, Heneghan H, Le Roux C, Pournaras DJ. Medication following bariatric surgery for type 2 diabetes mellitus (BY-PLUS) study: rationale and design of a randomised controlled study. BMJ Open. 2022 Jul 25;12(7):e054313. doi: 10.1136/bmjopen-2021-054313. PMID 35879015